CLINICAL TRIAL: NCT06247553
Title: To Develop a Walking Exercise Program for Non-ambulatory Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOD00042952
Record Dates: First submitted 2023-03-22; First posted 2024-02-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Walking, Difficulty; Cardiovascular Injury
Keywords: stroke; unable to walk
MeSH Terms: conditions — Stroke; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single-blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait Training (Experimental): The gait training in the experimental group will use a treadmill with a partial body-weight support system and our gait training device. A gait training session will include 2-minute warming up at the beginning and 2-minute cooling down at the end, at a treadmill speed of 0.6 mph. After the warming up, the treadmill speed will increase at every two minutes by an increment of 0.2 mph. Participant's heart rate will be monitored throughout the training session by using a Polar OH1 optical HR sensor placed in the participant's left forearm. Reseachers will stop the increase and maintain the same treadmill speed after the HR reaching the target heart rate zone of 50% - 60% of age-predicted heart rate reserve.
  Interventions: Other: Gait Training
- Leg Cycling Exercise (Active Comparator): The leg cycling exercise will use a stationary bicycle and the similar protocol as in the experimental group. The cycling exercise will include 2-minute warming up in the beginning and 2-minute cooling down at the end with a speed of 10 rpm and resistance of level 1 of 4. After warming up, the speed will increase at every two minutes by an increment of 5 rpm until reaching the target heart rate zone of 50% - 60% of age-predicted maximum heart rate. If the participant cannot tolerate any more increase in cycling speed before reaching the target heart rate, the resistance will be increased. The training duration will be individualized at the beginning and increase weekly by 5 minutes, depending on the tolerance of the participant, up to the maximum of 30 minutes. Both heart rate and blood pressure will be monitored before, during, and after each session to ensure safety. Each session including setting up will be about one hour.
  Interventions: Other: Leg Cycling Exercise

INTERVENTIONS:
Other: Gait Training — The gait training in the experimental group will use a treadmill with a partial body-weight support system and our gait training device. A gait training session will include 2-minute warming up at the beginning and 2-minute cooling down at the end, at a treadmill speed of 0.6 mph. After the warming up, the treadmill speed will increase at every two minutes by an increment of 0.2 mph. Participant's heart rate will be monitored throughout the training session by using a Polar OH1 optical HR sensor placed in the participant's left forearm. Researchers will stop the increase and maintain the same treadmill speed after the HR reaching the target heart rate zone of 50% - 60% of age-predicted heart rate reserve.
  Arms: Gait Training
Other: Leg Cycling Exercise — The leg cycling exercise will use a stationary bicycle and the similar protocol as in the experimental group. The cycling exercise will include 2-minute warming up in the beginning and 2-minute cooling down at the end with a speed of 10 rpm and resistance of level 1 of 4. After warming up, the speed will increase at every two minutes by an increment of 5 rpm until reaching the target heart rate zone of 50% - 60% of age-predicted maximum heart rate. If the participant cannot tolerate any more increase in cycling speed before reaching the target heart rate, the resistance will be increased. The training duration will be individualized at the beginning and increase weekly by 5 minutes, depending on the tolerance of the participant, up to the maximum of 30 minutes. Both heart rate and blood pressure will be monitored before, during, and after each session to ensure safety. Each session including setting up will be about one hour.
  Arms: Leg Cycling Exercise

SUMMARY:
The goal of this clinical trial is to test a gait (walking) training program in non-ambulatory (unable to walk) chronic stroke survivors. The main question it aims to answer is:

• Will gait training improve the cardiovascular system in non-ambulatory chronic stroke survivors better than a sitting leg cycling exercise?

Participants will walk on a treadmill with a partial body-weight support system and the gait training device. Researchers will compare with a leg-cycling exercise to see if there are significant differences in resting heart rate, systolic blood pressure (SBP), and A1c levels in the blood.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and permanent disability. About 795,000 strokes occur in the US each year and more than seven million Americans are living with effects of stroke. Cardiovascular diseases are commonly presented and are primary causes of death in stroke survivors. Numerous studies have proven the benefits of walking or other forms of aerobic exercise for cardiovascular and pulmonary function in people after stroke. This proposed randomized controlled efficacy trial will primarily examine whether the investigators' gait training can improve the cardiovascular system in non-ambulatory chronic stroke survivors better than a sitting leg cycling exercise. The investigators have recently developed a novel gait training device and a training program. The experimental group in the proposed project will undergo an 8-week gait training program using a treadmill with body-weight support and the investigators' novel gait training device. The control group will receive an 8-week sitting leg cycling exercise program with similar exercise intensity, frequency, and duration. The proposed project will examine differences between the two groups using a set of comprehensive outcome assessments of cardiovascular, pulmonary, and sensorimotor functions.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 to 80 years old
* male or female
* independent ambulation before stroke
* able to understand and follow verbal commands in English
* have physicians' approval for exercise
* be in a stable medical condition
* must be after the first stroke
* unable to walk independently
* in the chronic stage (at least 6 months after stroke onset)

Exclusion Criteria:

* musculoskeletal or other disorders that prevent the participant from participating in the exercise
* blood pressure higher than 200/110 mm Hg
* diagnosis of severe depression
* functionally restricted passive movement in the major joints of lower limbs
* unable to speak or understand English
* unable to travel to the Research Laboratory
* currently participate in other walking training using treadmill with or without a body-weight support system
* body weight greater than 400 lbs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
changes in resting heart rate (rHR) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  Resting heart rate (measured in beats per minute) will be measured using a Polar heart rate monitoring system.
systolic blood pressure (SBP) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  Systolic blood pressure (measured in mmHg) will be measured using a mercury sphygmomanometer.
glycated hemoglobin (HbA1c) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  HbA1c levels will be measured by collecting a drop of blood from the middle finger of the unaffected hand and use the A1CNow+ System for analysis.

SECONDARY OUTCOMES:
changes in diastolic blood pressure (DBP) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  Diastolic blood pressure (measured in mmHg) will be measured using a mercury sphygmomanometer.
changes in forced vital capacity (FVC) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  To obtain FVC measurements (measured in liters (L)) nose clip will be used, and subject's lips will be sealed around the mouthpiece to prevent air from leaking. The study team member will verbally encourage the subject to keep inhaling and exhaling at the maximum capacity. For FVC measurement, the subject will be instructed to maximally inhale, and immediately exhale forcibly and maximally. This test will be repeated at least three times. At least one minute will be allowed between each repetition to avoid fatigue.
clinical measurement of Functional Ambulation Category (FAC) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  The measurement of FAC will determine an individual's walking ability based on the amount of human assistance needed. It includes six categories, with Category 0 indicating nonfunctional ambulation and Category 5 - independent ambulation on varying surfaces.
changes in exercise heart rate (eHR) | These will be measured pre- and post-exercise for the intervention group.
  Heart rate will be obtained using a Polar heart rate monitoring system.
changes in low-density lipoprotein cholesterol (LDL-C) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  A blood sample will be drawn from the antecubital vein in the unaffected arm to be analyzed for plasma cholesterol (LDL-C) levels.
changes in vital capacity (VC) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  To obtain VC measurements (measured in liters (L)) nose clip will be used, and subject's lips will be sealed around the mouthpiece to prevent air from leaking. The study team member will verbally encourage the subject to keep inhaling and exhaling at the maximum capacity. The subject will sit and first be asked to breathe normally three times. The subject will then be instructed immediately to maximally inhale or exhale and repeat four times. This test will be repeated at least three times. At least one minute will be allowed between each repetition to avoid fatigue.
changes in Berg Balance Scale (BBS) score | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  The BBS is a test consisting of 14 items, designed to measure balance performance in sitting, standing, and weight transfer activities. The minimum score is 0 and the maximum score is 56. Higher scores indicate greater balance performance.
changes in muscle activity of the affected leg for participants in the intervention group | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  The muscle activity will be measured by the recorded muscle electromyogram (EMG) signals.
changes in heart rate variability (HRV) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  Heart rate variability will be obtained using electrocardiography (ECG).
changes in stroke volume (SV) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  Stroke Volume (SV), an indication of cardiac functioning, will be measured by non-invasive impedance cardiography.
changes in cardiac output (CO) | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.
  Cardiac Output (CO), an indication of cardiac functioning, will be measured by non-invasive impedance cardiography.

OTHER OUTCOMES:
changes in PASS, Postural Assessment Scale for Stroke Patients | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The PASS has 12 items that assess balancing ability. The minimum score is 0 and the maximum score is 36. Higher scores indicate greater balancing ability.
changes in TIS, Trunk Impairment Scale | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The TIS has 17 items that assess trunk functionality and impairment. The minimum score is 0 and the maximum score is 23. Higher scores indicate greater trunk functionality and less impairment.
changes in MI, Motricity Index | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The MI has 6 items (repeated for each arm and leg) that assess motor impairment in stroke patients.
changes in RNLI, Reintegration to Normal Living Index | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The RNLI has 11 items to assess the extent of the patient's ability to return to normal living activities.
changes in MBI, Modified Barthel Index | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The MBI has 11 items assessing patients' ability complete a variety of self-care tasks.
changes in HADS, Hospital Anxiety and Depression Scale | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The HADS has 14 items (7 depression items and 7 anxiety items) to assess depression and anxiety symptoms experienced in the past week. The minimum score is 0 and the maximum score is 21 for depression and anxiety individuals. Higher scores on depression items indicate higher depression. Higher scores on anxiety items indicate higher anxiety.
MoCA, Montreal Cognitive Assessment | All participants will be assessed at baseline (during the evaluation).
  The MoCA has 8 items that assess cognitive functioning.
BMI, Body Mass Index | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  BMI will be measured by obtaining height and weight.
changes in walking endurance and capacity | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  Walking endurance and capacity will be measured with the total distance covered when performing a 6-minute overground walking test involving walking as far as possible for 6 minutes on a flat, marked course.
changes in walking speed, joint motion, and muscle activation | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  Walking speed, joint motion, and muscle activation will be measured when performing a 6-meter overground walking test involving walking a 6-meter distance on a flat, marked course.
Modified Functional Reach Test | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The modified functional reach test assess balance by measuring reaching ability 3 times under 3 conditions to assess balance.
Fugl Meyer Lower Extremity | All participants will be assessed at baseline (during the evaluation) and at the end of the 8-week intervention.]
  The Fugl Meyer Lower Extremity assessment assesses impairment in motor function, balance, sensation and joint functioning with 43 items.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No